CLINICAL TRIAL: NCT05570032
Title: Effectiveness of Virtual Reality Training in Gait Improvement of Post Stroke Patients: A Quasi-experimental Study
Brief Title: Effectiveness of Virtual Reality Training in Gait Improvement of Post Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Hazrat Bilal PT (Other)
Responsible Party: Sponsor-Investigator, Dr. Hazrat Bilal PT, Co-Invistigator, NCS University System
Organization: NCS University System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMU/IPMR/VR
Record Dates: First submitted 2022-09-26; First posted 2022-10-06 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual reality training (Experimental): In intervention the participants took part in the VR training. The X-BOX 360 (Augmented virtual reality) device was used. The participants were guided about the virtual reality training including Kinect sports gamming (Trail 1. badminton, beach volley ball, Soccer goal keeping). Each training was performed for 15 minutes with 5 minutes break time. The whole training was performed for 8 weeks. After eight weeks final assessment was done through outcome measuring tools (TUG test, MAS scale, forward stepping test and Functional reach test).
  Interventions: Device: Virtual Reality Training

INTERVENTIONS:
Device: Virtual Reality Training — In intervention the participants took part in the VR training. The X-BOX 360 (Augmented virtual reality) device was used. The participants were guided about the virtual reality training including Kinect sports gamming (Trail 1. badminton, beach volley ball, Soccer goal keeping). Each training was performed for 15 minutes with 5 minutes break time. The whole training was performed for 8 weeks. After eight weeks final assessment was done through outcome measuring tools (TUG test, MAS scale, forward stepping test and Functional reach test).

SUMMARY:
This single group quasi-experimental study was conducted at Rafsan Neuro Rehab Center, Peshawar from October 2021 to February 2022. The sample size of study was 40 post stroke patients who were diagnosed on physical findings and other investigation like CT and MRI. The inclusion criteria were set as post-stroke patients for more than 3 months with 20 and above score on MAS scale and age of 55 to 65 years, while the exclusion criteria were defined as participants having traumatic brain injuries, degenerative brain diseases, post craniotomy tumor patients leading to hemiplegia, patients having recurrent episodes of stroke, stroke patient with dementia and score on MAS scale below 20.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were set as post-stroke patients for more than 3 months
* 20 and above score on MAS scale
* age of 55 to 65 years

Exclusion Criteria:

* The exclusion criteria were defined as
* participants having traumatic brain injuries, degenerative brain diseases, post craniotomy tumor patients leading to hemiplegia,
* patients having recurrent episodes of stroke,
* stroke patient with dementia
* score on MAS scale below 20.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
TUG test | 8 weeks
  Objective of the TUG test is to determine fall risk and measure the progress of balance, sit to stand and walking.
MAS scale | 8 weeks
  The Motor Assessment Scale (MAS) is a performance-based scale used to assess level of impairment and everyday motor function in patients with stroke.
Forward stepping test | 8 weeks
  Forward stepping test is used to assess the balance of the patients with stroke or other neurological disorder.
Functional reach test | 8 weeks
  The Functional reach test assesses a patient's stability by measuring the maximum distance an individual can reach forward while standing in a fixed position.

CONTACTS AND LOCATIONS:
Overall Officials: Shakir Ullah, MSPT, Principal Investigator — Khyber Medical University Peshawar
Locations (1):
- Hazrat Bilal, Peshawar, Khyber Pakhtunkhwa, Pakistan